CLINICAL TRIAL: NCT05086679
Title: Compression Stockings for Treating Vasovagal Syncope (COMFORTS II) Trial; a Double Blind, Multi-center Randomized Controlled Trial
Brief Title: Compression Stockings for Treating Vasovagal Syncope Trial
Acronym: COMFORTS II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran Heart Center (Other)
Collaborators: Tehran Arrhythmia Center (Unknown); Rajaie Cardiovascular Medical and Research Center (Other); Imam Khomeini Hospital (Other); Isfahan University of Medical Sciences (Other); Ahvaz Jundishapur University of Medical Sciences (Other); Guilan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masih Tajdini, MD, Associate Professor of Cardiology, Tehran Heart Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1400-2-101-54781
Record Dates: First submitted 2021-10-05; First posted 2021-10-21 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Syncope, Vasovagal
Keywords: Syncope, Vasovagal; Syncope; Compression stocking; Randomized Clinical Trial
MeSH Terms: conditions — Syncope, Vasovagal; Syncope | interventions — Stockings, Compression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression stockings with 25-30 mm Hg pressure (Active Comparator): Compression stockings with 25-30 mm Hg pressure, as long as they could (ideal would be the majority of the time they are upright)
  Interventions: Device: Compression Stockings with 25-30 mm Hg pressure; Behavioral: Lifestyle modification
- Compression stockings with up to 10 mm Hg pressure (Sham Comparator): Compression stockings with up to <=10 mm Hg pressure, as long as they could (ideal would be the majority of the time they are upright)
  Interventions: Device: Compression stockings with up to <=10 mm Hg pressure; Behavioral: Lifestyle modification

INTERVENTIONS:
Device: Compression Stockings with 25-30 mm Hg pressure — The group will have compression stockings with 25-30 mm Hg pressure. All the participants' size for compression stocking will be measured at the first visit. Three points will be measured: below and above their knees and above their ankle. Subsequently, Right Arian Farmed Co (Tehran, Iran) will provide compression stockings for patients based on their sizes. Participants will be asked to use compression stockings as long as they could (ideal would be the majority of the time they are upright). In addition, a CD included some videos and booklets about instructions on how to wear CS and how to keep them will be provided for the participants with their compression stockings.
  Arms: Compression stockings with 25-30 mm Hg pressure
Device: Compression stockings with up to <=10 mm Hg pressure — The group will have compression stockings with up to 10 mm Hg pressure. All the participants' size for compression stocking will be measured at the first visit. Three points will be measured: below and above their knees and above their ankle. Subsequently, Right Arian Farmed Co (Tehran, Iran) will provide compression stockings for patients based on their sizes. Participants will be asked to use compression stockings as long as they could (ideal would be the majority of the time they are upright). In addition, a CD included some videos and booklets about instructions on how to wear CS and how to keep them will be provided for the participants with their compression stockings.
  Arms: Compression stockings with up to 10 mm Hg pressure
Behavioral: Lifestyle modification — All patients will receive standard treatment of VVS despite their randomization(drink 2-3 liters of fluids, consume 10 grams 120 mmol/day of sodium chloride, and practice counter-pressure maneuvers (squatting, leg crossing, handgrip, and arm-tensing))

SUMMARY:
Syncope, a sudden, transient loss of consciousness (TLOC), is a common inconvenience of daily function and quality of life (QoL). The vasovagal syncope (VVS) is the most common type of syncope, which central and peripheral stimuli may trigger syncope by decreasing peripheral vascular resistance, bradycardia, or both. The venous return to the heart is one of these triggers which its reduction may occur due to prolonged standing, hot environment, hypovolemia, or redistribution of blood volume. The compression stockings may reduce syncopal episodes by increasing venous return. Although the use of compression stockings was never assessed in clinical trials, it could be a possible treatment for decreasing VVS recurrences.

DETAILED DESCRIPTION:
The COMFORTS II study is designed as a multicenter, longitudinal, double blind, parallel design RCT to assess the beneficial effect of compression stockings for preventing recurrences of VVS. The participants will be treated by the standard treatment of VVS, and then they will be randomized into two groups (1:1 ratio) to use compression stockings, one group with 25-30 mm Hg pressure and the other one with <= 10 mmHg pressure, Randomization and allocation concealment will be done by the primary investigators (www.comfortstrial.com). To balance participant enrolment, participating centers will stratify the randomization block. The enrolling physicians will be blinded to the randomization to minimize the selection bias. Hence, the randomization code will not be revealed till the patient has been enrolled, and the baseline features and consent form have been uploaded.

The syncope Unit of Tehran Heart Center (SUTHC), Tehran University of Medical Sciences is the primary investigation site (same as COMFORTS I trial). Seven study centers across Iran declared their commitment to participate in this study. After randomization, participants will be allocated their treatment as one group will have compression stockings with 25-30 mm Hg pressure and in the control group pressure will be limited up to <=10 mmHg, which elastic compression stockings will be sent to patients by post. Participants will be asked to use compression stockings as long as they could (ideal would be the majority of the time they are upright). Adherence of patients to the use of compression stockings will be daily with predefined forms given to patients after randomization. In addition, a CD included some videos and booklets about instructions on how to wear CS and how to keep them will be provided for the participants with their compression stockings. All patients will receive standard treatment of VVS despite their randomization. According to syncope guidelines, patients will learn to drink 2-3 liters of fluids, consume 10 grams 120 mmol/day of sodium chloride, and practice counter-pressure maneuvers (squatting, leg crossing, handgrip, and arm-tensing

After six months of follow-up for 50% of the study participants, event rates will be assessed by the data and safety monitoring board (DSMB) and the sample size can be adjusted based on DSMB guidance

Data safety and monitoring board (DSMB):

a. Roles: i. Monitoring data quality and completeness, as well as timeliness of enrollment, visit, and follow-up, ii. Overseeing adherence to trial protocol and providing feedback in documented reports to the trial committee iii. Overseeing performance of individual centers, and providing feedback in documented reports to the trial committee iv. Monitoring patient safety and their current treatment, and recommending changes in therapies for individuals subjects if needed, v. Advising adjustments to the sample size after interim analysis of data upon completion of six months of follow-up for half of the study sample size, vi. Monitoring scientific or therapeutic developments in the field, and in case of major developments providing updated recommendations on the ethics of the study.

b. Meetings: i. At the start of enrollment ii. Every three months after beginning of enrollment until the final follow-up iii. After formal analysis of the data has been performed iv. The chair of DSMB may call for additional meetings

c. Members: i. Chair: Dr. Haleh Ashraf (Sina Hospital); The chair of DSMB is responsible for conducting meetings, and may add members to the DSMB at her own discretion. ii. Mohammad-Reza Malekpour (Non-communicable Diseases Research Center, Endocrinology and Metabolism Population Sciences Institute) iii. Maryam Masoudi (Roozbeh Psychiatric Hospital)

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18≤age≤65
* VVS as the cause of TLOC confirmed by Clinical diagnosis And CSSS ≥-2
* ≥2 episodes of VVS during the last year
* The capability of giving informed consent
* Signed written informed consent

Exclusion Criteria:

* Orthostatic hypotension (decrease in BP ≥20/10 mmHg after 5-minute stand test)
* Postural tachycardia (increase in heart rate ≥30 bpm after 5-minute stand test)
* Carotid sinus hypersensitivity (ventricular pause >3 or decrease in BP > 50 mmHG after carotid sinus massage, performed in patients 40 years or older)
* History of Seizure
* Currently using midodrine or fludrocortisone
* Cardiac rhythm disorders including ventricular tachycardia, long QT syndrome, Brugada syndrome, ARVC, CHB, or any conduction abnormality on ECG
* Severe valvular heart disease
* Hypertrophic cardiomyopathy
* Cardiac systolic dysfunction (ejection fraction ≤40%)
* Obstructive coronary artery disease
* Cardiac implantable electronic devices
* Prior recommendation of ECS by a health-care provider, or other indication for ECS use
* Foot ulcers and diabetic foot
* Chronic venous insufficiency
* Renal failure stage ≥3 (eGFR <60 mL/min/1.73 m2)
* Presence of a chronic severe illness
* Pregnancy, or intention to become pregnant in the next year
* Unwillingness to participate or to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with recurrence of VVS | The follow-up continues for 12 months after randomization
  The proportion of participants with recurrence of VVS to all participants in their arm of treatment during the follow-up
The time to the first syncopal episode | The follow-up continues for 12 months after randomization
  Time from randomization to occurrence of the first episode of vasovagal syncope during the follow-up

SECONDARY OUTCOMES:
The frequency of syncopal episodes | The follow-up continues for 12 months after randomization
  The frequency of syncopal episodes in the follow-up period
The time intervals between recurrent episodes | The follow-up continues for 12 months after randomization
  The time between recurrent episodes of syncope
Patient-reported adverse events | The follow-up continues for 12 months after randomization
  Patient-reported adverse events in the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Hamed Tavolinejad, MD, Study Director — Tehran Heart Center, Tehran University of Medical Sciences; Amirhossein Poopak, MD, Study Director — Tehran Heart Center, Tehran University of Medical Sciences
Locations (1):
- Tehran Heart Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
The data is not publicly available due to privacy/ethical restrictions. The data can be shared upon reasonable request to the trial committee.

REFERENCES:
- [Background] Sadeghian S, Aminorroaya A, Tajdini M. The Syncope Unit of Tehran Heart Center. Eur Heart J. 2021 Jan 7;42(2):148-150. doi: 10.1093/eurheartj/ehaa532. No abstract available. PMID 33346809
- [Background] Aminorroaya A, Tavolinejad H, Sadeghian S, Jalali A, Alaeddini F, Emkanjoo Z, Mollazadeh R, Bozorgi A, Oraii S, Kiarsi M, Shahabi J, Akbarzadeh MA, Rahimi B, Joharimoghadam A, Mohsenizade A, Mohammadi R, Oraii A, Ariannejad H, Apakuppakul S, Ngarmukos T, Tajdini M. Comparison of Outcomes with Midodrine and Fludrocortisone for Objective Recurrence in Treating Syncope (COMFORTS trial): Rationale and design for a multi-center randomized controlled trial. Am Heart J. 2021 Jul;237:5-12. doi: 10.1016/j.ahj.2021.03.002. Epub 2021 Mar 6. PMID 33689731